CLINICAL TRIAL: NCT01298141
Title: A Multicenter Open-Label Treatment Protocol to Observe the Safety of Replagal® (Agalsidase Alfa) Enzyme Replacement Therapy in Canadian Patients With Fabry Disease
Brief Title: A Multicenter Open-Label Treatment Protocol to Observe the Safety of Replagal (Agalsidase Alfa) Enzyme Replacement Therapy in Canadian Patients With Fabry Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGT-REP-081
Record Dates: First submitted 2011-02-15; First posted 2011-02-17 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Fabry Disease
Keywords: Replagal; Enzyme Replacement Therapy; agalsidase alfa
MeSH Terms: conditions — Fabry Disease | interventions — agalsidase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Replagal® (Experimental): All eligible patients may receive Replagal produced by the bioreactor process (AF Replagal) on this treatment plan until AF Replagal is commercially available for the patient, the patient's participation is discontinued, or the study is discontinued, whichever comes first.
  Interventions: Biological: agalsidase alfa

INTERVENTIONS:
Biological: agalsidase alfa — Cohort 1: 0.2 mg/kg body weight administered as an intravenous (IV) infusion over 40 minutes every other week (EOW)
  Cohort 2: 0.2 mg/kg body weight administered as an intravenous (IV) infusion over 40 minutes weekly
  Other Names: Replagal

SUMMARY:
The purpose of this study is to observe the safety of agalsidase alfa in Canadian patients with Fabry disease.

DETAILED DESCRIPTION:
This study will evaluate the safety of agalsidase alfa in patients with Fabry disease.

Patients diagnosed with Fabry disease who meet current Canadian guidelines for enzyme replacement therapy will be eligible to enroll in the study and will receive agalsidase alfa at a dose of 0.2 mg/kg body weight administered by an IV infusion over 40 minutes every week or every other week, based on previous treatment.

Shire has implemented a change to the drug substance manufacturing process. Safety data will be collected in patients receiving product manufactured with this process. There are no changes to the drug product formulation, manufacturing site, manufacturing process, and container closure.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1:

1. The patient has a documented diagnosis of Fabry disease.
2. The patient is sufficiently compliant with study activities to participate in this treatment plan, as judged by the Investigator.
3. The patient must meet current Canadian guidelines for enzyme replacement therapy for Fabry disease by meeting one of the following criteria:

   1. Age-adjusted glomerular filtration rate (GFR) <80 ml/min or a decline in GFR of >10% which is sustained for 3 months and for which other causes of declining renal function have been excluded by a nephrologist or any 2 of the following:

      * Isolated proteinuria ≥500 mg/day/1.73 m2 without other cause
      * Nephrogenic diabetes insipidus
      * Fanconi syndrome
      * Hypertension
   2. Evidence of cardiac involvement related to Fabry disease including any 2 of the following:

      * Left ventricular (LV) wall thickness >12 mm
      * Left ventricular hypertrophy (LVH) by electrocardiogram (ECG); Estes ECG score must be >5
      * Left ventricular mass index (LVMI) by 2D echocardiogram 20% above normal for age
      * Diastolic filling abnormalities by 2D echocardiogram or by other accepted measures of diastolic filling. E/A ration >2.0 and deceleration time <140 msec
      * Increase of LV mass of at least 5 g/m2/year, with three measurements over a minimum of 12 months
      * Increase of left atrium (LA) size on 2D echo at least 10% above normal for age. In parasternal long axis view (PLAX) >33 mm; in four chamber view >42 mm
      * Cardiac conduction and rhythm abnormalities: atrioventricular (AV) block, short PR interval, left branch bundle block (LBBB), ventricular or atrial tachyarrhythmias, sinus bradycardia (in the absence of drugs with negative chronotropic activity)
      * Delayed posterolateral left ventricular wall late enhancement on MRI as evidence of advanced cardiac disease with fibrosis
   3. Evidence of neurological involvement related to Fabry disease including 1 of the following:

      * Stroke or transient ischemic attack (TIA) prior to the age of 55 documented by a neurologist
      * Acute onset unilateral hearing loss
      * Acut monocular visual loss without other cause
   4. Chronic, intractable diarrhea and/or abdominal pain/cramps, refractory to standard management for at least 6 months.
   5. Chronic, intractable neuropathic pain, refractory to analgesics and standard pain management for at least 6 months.

   Cohort 2:
4. Patient must have participated in Study REP001a.

Exclusion Criteria:

1. The patient has experienced an anaphylactic or anaphylactoid reaction or other infusion-related reaction which, in the opinion of the Investigator, precludes further treatment with agalsidase alfa or may interfere with the interpretation of the study.
2. The patient is otherwise unsuitable for the study, in the opinion of the Investigator.
3. The patient is enrolled in another clinical study, other than the Canadian Fabry Disease Initiative (CFDI).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2011-08-10 (Actual); Primary Completion 2017-09-25 (Actual); Study Completion 2017-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (12):
- Canada (12):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Izaak Walton Killam (IWK) Health Centre, Halifax, Nova Scotia
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre - Victoria Hospital, London, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - The Fred A. Litwin Family Centre in Genetic Medicine, Toronto, Ontario
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke (CHUS), Sherbrooke, Quebec

REFERENCES:
- [Derived] Khan A, Sirrs SM, Bichet DG, Morel CF, Tocoian A, Lan L, West ML; Canadian Fabry Disease Initiative. The Safety of Agalsidase Alfa Enzyme Replacement Therapy in Canadian Patients with Fabry Disease Following Implementation of a Bioreactor Process. Drugs R D. 2021 Dec;21(4):385-397. doi: 10.1007/s40268-021-00361-4. Epub 2021 Sep 20. PMID 34542871

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted at 12 sites in Canada between 10 Aug 2011 (first participant first visit) and 25 Sep 2017 (last participant last visit).
Pre-assignment Details: A total of 171 participants enrolled into cohort 1 (participants from Canadian Fabry Disease Initiative [CFDI]) and cohort 2 (participants who participated in study REP001a) and among them 167 participants received at least one full or partial dose of Replagal (agalsidase alfa) animal free (AF).
Groups:
- Replagal (Agalsidase Alfa): Participants in cohort 1 received Replagal AF intravenous (IV) infusion at a dose of 0.2 milligram per kilogram (mg/kg) body weight every other week (EOW) and cohort 2 received Replagal AF IV infusion at a dose of 0.2 mg/kg body weight weekly until the drug became commercially available or the participant discontinued, whichever came first.
Period: Overall Study
Arm/Group | Replagal (Agalsidase Alfa)
Started | 171
Treated | 167
Completed | 140
Not Completed | 31
Not completed — Adverse Event | 3
Not completed — Refusal of Required Study Procedures | 1
Not completed — Withdrawal by Subject | 6
Not completed — Termination of Study by the Investigator | 5
Not completed — Other | 5
Not completed — Lost to Follow-up | 1
Not completed — Death | 6
Not completed — Not treated | 4

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received at least one full or partial infusion of Replagal AF.
Groups:
- Replagal (Agalsidase Alfa): Participants in cohort 1 received Replagal AF IV infusion at a dose of 0.2 mg/kg body weight EOW and cohort 2 received Replagal AF IV infusion at a dose of 0.2 mg/kg body weight weekly until the drug became commercially available or the participant discontinued, whichever came first.
Arm/Group | Replagal (Agalsidase Alfa)
Number analyzed (Participants) | 167
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at Informed Consent
  Years | 48.85 (14.821)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 165
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 160
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any noxious, pathologic, or unintended change in anatomical, physiologic, or metabolic function as indicated by physical signs, symptoms, or laboratory changes occurring in any phase of a clinical study, whether or not considered investigational product-related.Treatment-emergent adverse events (TEAEs) were defined as those events which occurred or worsened in severity after first treatment with Replagal AF until 30 days after the last dose. A serious AE (SAE) was any AE occurred at any dose that resulted in death, life-threatening, hospitalization, prolongation of existing hospitalization, persistent or significant disability or incapacity and congenital anomaly or birth defect.
Time Frame: From the start of study treatment up to 30 days after the last dose of study drug administration (up to 320 weeks)
Population: Safety Population included all participants who received at least one full or partial infusion of Replagal AF.
Measure: Count of Participants; unit: Participants
Arm/Group | Replagal (Agalsidase Alfa)
Number analyzed (Participants) | 167
Participants
  Any TEAE | 163
  Any Serious TEAE | 74
  Any TEAE Leading to Treatment Discontinuation | 7

2. Primary Outcome: Number of Participants With Infusion-Related Reactions (IRR)
Description: An IRR (also referred to as infusion-related adverse event [IRAE]) was defined as an AE that began either during the infusion or within 12 hours after the start of the infusion and was judged as possibly or probably related to study drug. The IRRs were classified based on the severity as Mild=No limitation of usual activities, Moderate=Some limitation of usual activities, Severe=Inability to carry out usual activities and Life-threatening=Immediate risk of death. The number of participants with infusion-related reactions was reported.
Time Frame: From the start of study treatment up to 30 days after the last dose of study drug administration (up to 320 weeks)
Population: Safety Population included all participants who received at least one full or partial infusion of Replagal AF.
Measure: Count of Participants; unit: Participants
Arm/Group | Replagal (Agalsidase Alfa)
Number analyzed (Participants) | 167
Participants
  Mild | 21
  Moderate | 16
  Severe | 3
  Life-threatening | 0

3. Primary Outcome: Number of Participants Who Reported Positive to Immunoglobulin A (IgA)
Description: The IgA status was measured using enzyme-linked immunosorbent assay (ELISA). Number of participants who reported positive to IgA was reported.
Time Frame: Baseline (within 6 months prior to first dose) up to Week 129
Population: Safety population included all participants who received at least one full or partial infusion of Replagal AF.
Measure: Count of Participants; unit: Participants
Arm/Group | Replagal (Agalsidase Alfa)
Number analyzed (Participants) | 167
Participants | 10

4. Primary Outcome: Number of Participants Who Reported Positive to Immunoglobulin E (IgE)
Description: The IgE status was measured using ELISA. Number of participants who reported positive to IgE was reported.
Time Frame: Baseline (within 6 months prior to first dose) up to Week 129
Population: Safety population included all participants who received at least one full or partial infusion of Replagal AF.
Measure: Count of Participants; unit: Participants
Arm/Group | Replagal (Agalsidase Alfa)
Number analyzed (Participants) | 167
Participants | 1

5. Primary Outcome: Number of Participants Who Reported Positive to Immunoglobulin M (IgM)
Description: The IgM status was measured using ELISA. Number of participants who reported positive to IgM was reported.
Time Frame: Baseline (within 6 months prior to first dose) up to Week 129
Population: Safety population included all participants who received at least one full or partial infusion of Replagal AF.
Measure: Count of Participants; unit: Participants
Arm/Group | Replagal (Agalsidase Alfa)
Number analyzed (Participants) | 167
Participants | 48

6. Primary Outcome: Number of Participants Who Reported Positive to Anti-drug Antibody (ADA)
Description: The ADA status was measured using ELISA and electrochemiluminescent (ECL) immunoassay. Number of participants who reported positive to ADA was reported.
Time Frame: Baseline (within 6 months prior to first dose) up to Week 285
Population: Safety population included all participants who received at least one full or partial infusion of Replagal AF.
Measure: Count of Participants; unit: Participants
Arm/Group | Replagal (Agalsidase Alfa)
Number analyzed (Participants) | 167
Participants | 42

7. Primary Outcome: Number of Participants Who Reported Positive to Neutralizing Antibody (NAb)
Description: The NAb status was measured using enzyme activity inhibition assay. Number of participants who reported positive to NAb was reported.
Time Frame: Baseline (within 6 months prior to first dose) up to Week 285
Population: Safety population included all participants who received at least one full or partial infusion of Replagal AF.
Measure: Count of Participants; unit: Participants
Arm/Group | Replagal (Agalsidase Alfa)
Number analyzed (Participants) | 167
Participants | 27

ADVERSE EVENTS:
Time Frame: From the start of study treatment up to 30 days after the last dose of study drug administration (up to 320 weeks)
Arm/Group | Replagal (Agalsidase Alfa)
All-Cause Mortality (participants affected / at risk) | 6/167
Serious Adverse Events (participants affected / at risk) | 74/167
Other Adverse Events (participants affected / at risk) | 160/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Replagal (Agalsidase Alfa) (N=167)
Anaemia (Blood and lymphatic system disorders) | 5 (5)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Splenic neoplasm malignancy unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1)
Eye swelling (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (4)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 2 (3)
Paraesthesia oral (Gastrointestinal disorders) | 2 (2)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1)
Swollen tongue (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Device malfunction (General disorders) | 1 (1)
Malaise (General disorders) | 2 (2)
Non-Cardiac chest pain (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 2 (2)
Pyrexia (General disorders) | 2 (2)
Fabry's disease (Congenital, familial and genetic disorders) | 3 (3)
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 (2)
Acute coronary syndrome (Cardiac disorders) | 4 (4)
Acute myocardial infarction (Cardiac disorders) | 3 (3)
Angina pectoris (Cardiac disorders) | 6 (6)
Angina unstable (Cardiac disorders) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 5 (7)
Atrial flutter (Cardiac disorders) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 4 (4)
Coronary artery disease (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Hypertrophic cardiomyopathy (Cardiac disorders) | 2 (2)
Intracardiac thrombus (Cardiac disorders) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 7 (8)
Palpitations (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 7 (7)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Kidney transplant rejection (Immune system disorders) | 1 (2)
Bacteraemia (Infections and infestations) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1)
Beta haemolytic streptococcal infection (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 7 (9)
Cholangitis suppurative (Infections and infestations) | 1 (1)
Cytomegalovirus viraemia (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 2 (2)
Escherichia bacteraemia (Infections and infestations) | 2 (2)
Infection (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 1 (1)
Perihepatic abscess (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 7 (7)
Pneumonia adenoviral (Infections and infestations) | 1 (1)
Pneumonia cytomegaloviral (Infections and infestations) | 1 (1)
Pneumonia primary atypical (Infections and infestations) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Septic shock (Infections and infestations) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (4)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1)
Psychosis postoperative (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1)
Electrocardiogram qt prolonged (Investigations) | 1 (1)
Enterococcus test positive (Investigations) | 1 (1)
Heart rate decreased (Investigations) | 1 (1)
Troponin increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Nephropathy (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 7 (8)
Renal failure chronic (Renal and urinary disorders) | 8 (9)
Biloma (Hepatobiliary disorders) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 8 (8)
Hypoaesthesia (Nervous system disorders) | 1 (5)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 3 (3)
Tension headache (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 3 (4)
Tremor (Nervous system disorders) | 1 (1)
Aortic valve replacement (Surgical and medical procedures) | 1 (1)
Cardiac ablation (Surgical and medical procedures) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 (1)
Cardiac pacemaker replacement (Surgical and medical procedures) | 1 (1)
Cardiac pacemaker revision (Surgical and medical procedures) | 1 (1)
Implantable defibrillator insertion (Surgical and medical procedures) | 1 (1)
Implantable defibrillator replacement (Surgical and medical procedures) | 1 (1)
Mitral valve replacement (Surgical and medical procedures) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1)
Priapism (Reproductive system and breast disorders) | 1 (1)
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1 (1)
Piloerection (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Replagal (Agalsidase Alfa) (N=167)
Anaemia (Blood and lymphatic system disorders) | 11 (25)
Arthralgia (Musculoskeletal and connective tissue disorders) | 45 (68)
Back pain (Musculoskeletal and connective tissue disorders) | 46 (63)
Joint swelling (Musculoskeletal and connective tissue disorders) | 14 (17)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 22 (30)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 10 (12)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 23 (29)
Myalgia (Musculoskeletal and connective tissue disorders) | 21 (22)
Neck pain (Musculoskeletal and connective tissue disorders) | 14 (14)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 12 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 34 (49)
Flushing (Vascular disorders) | 9 (49)
Hypertension (Vascular disorders) | 17 (22)
Hypotension (Vascular disorders) | 17 (23)
Ear pain (Ear and labyrinth disorders) | 11 (11)
Tinnitus (Ear and labyrinth disorders) | 17 (17)
Vertigo (Ear and labyrinth disorders) | 23 (26)
Vision blurred (Eye disorders) | 16 (19)
Abdominal discomfort (Gastrointestinal disorders) | 13 (14)
Abdominal pain (Gastrointestinal disorders) | 29 (50)
Abdominal pain upper (Gastrointestinal disorders) | 17 (21)
Constipation (Gastrointestinal disorders) | 14 (16)
Diarrhoea (Gastrointestinal disorders) | 51 (90)
Dyspepsia (Gastrointestinal disorders) | 11 (12)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 11 (12)
Haematochezia (Gastrointestinal disorders) | 9 (9)
Nausea (Gastrointestinal disorders) | 57 (119)
Vomiting (Gastrointestinal disorders) | 44 (79)
Asthenia (General disorders) | 14 (18)
Chest discomfort (General disorders) | 11 (16)
Chest pain (General disorders) | 16 (22)
Chills (General disorders) | 15 (30)
Fatigue (General disorders) | 70 (95)
Influenza like illness (General disorders) | 14 (21)
Non-Cardiac chest pain (General disorders) | 23 (27)
Oedema (General disorders) | 9 (10)
Oedema peripheral (General disorders) | 56 (82)
Pain (General disorders) | 16 (21)
Pyrexia (General disorders) | 28 (35)
Angina pectoris (Cardiac disorders) | 22 (44)
Palpitations (Cardiac disorders) | 35 (49)
Bronchitis (Infections and infestations) | 18 (21)
Cellulitis (Infections and infestations) | 11 (15)
Cystitis (Infections and infestations) | 11 (15)
Ear infection (Infections and infestations) | 13 (14)
Influenza (Infections and infestations) | 31 (45)
Localised infection (Infections and infestations) | 12 (17)
Lower respiratory tract infection (Infections and infestations) | 19 (21)
Nasopharyngitis (Infections and infestations) | 64 (123)
Pneumonia (Infections and infestations) | 11 (18)
Sinusitis (Infections and infestations) | 17 (25)
Upper respiratory tract infection (Infections and infestations) | 14 (20)
Urinary tract infection (Infections and infestations) | 23 (38)
Contusion (Injury, poisoning and procedural complications) | 21 (29)
Skin laceration (Injury, poisoning and procedural complications) | 9 (10)
Cardiac murmur (Investigations) | 12 (16)
Temperature difference of extremities (Investigations) | 16 (18)
Gout (Metabolism and nutrition disorders) | 9 (16)
Balance disorder (Nervous system disorders) | 9 (9)
Dizziness (Nervous system disorders) | 54 (85)
Headache (Nervous system disorders) | 54 (104)
Hypoaesthesia (Nervous system disorders) | 26 (31)
Migraine (Nervous system disorders) | 13 (16)
Neuralgia (Nervous system disorders) | 32 (63)
Paraesthesia (Nervous system disorders) | 29 (31)
Syncope (Nervous system disorders) | 10 (11)
Tremor (Nervous system disorders) | 17 (19)
Anxiety (Psychiatric disorders) | 19 (22)
Depression (Psychiatric disorders) | 12 (13)
Insomnia (Psychiatric disorders) | 13 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 51 (82)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 40 (58)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 14 (16)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 (25)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 16 (19)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 24 (34)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 11 (17)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 10 (11)
Angiokeratoma (Skin and subcutaneous tissue disorders) | 11 (11)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 19 (29)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (13)
Rash (Skin and subcutaneous tissue disorders) | 18 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (7):
  • Study Protocol: Original Protocol (2010-09-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT01298141/Prot_000.pdf
  • Study Protocol: Amendment 1 (2010-11-23): https://cdn.clinicaltrials.gov/large-docs/41/NCT01298141/Prot_001.pdf
  • Study Protocol: Amendment 2 (2010-12-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT01298141/Prot_002.pdf
  • Study Protocol: Amendment 3 (2011-09-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT01298141/Prot_003.pdf
  • Study Protocol: Amendment 4 (2013-03-28): https://cdn.clinicaltrials.gov/large-docs/41/NCT01298141/Prot_004.pdf
  • Study Protocol: Amendment 5 (2015-03-27): https://cdn.clinicaltrials.gov/large-docs/41/NCT01298141/Prot_005.pdf
  • Statistical Analysis Plan (2017-12-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT01298141/SAP_006.pdf